CLINICAL TRIAL: NCT02730572
Title: Concerta-to-Generic Switch Study
Brief Title: Concerta (Methylphenidate) -To-Generic Switch Study
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107709; RRA 14797 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concerta to authorized generic (AG) formulation: Participants in the Truven Commercial Claims and Encounters (CCAE) database who enroll in the study will have a confirmed diagnosis of ADHD and continuously using Concerta for at least 60 days. Participants who will switch from Concerta to AG formulation will be observed.
  Interventions: Drug: Concerta; Drug: Concerta AG formulation
- Concerta to equivalent generic (EG) formulation: Participants in the Truven Commercial Claims and Encounters (CCAE) database who enroll in the study will have a confirmed diagnosis of ADHD and continuously using Concerta for at least 60 days. Participants who will switch from Concerta to EG formulation will be observed.
  Interventions: Drug: Concerta; Drug: Concerta EG formulation

INTERVENTIONS:
Drug: Concerta — This is an observational study. Participants who have been on Concerta for at least 60 days will be observed.
  Other Names: Methylphenidate
Drug: Concerta AG formulation — This is an observational study. Participants who have been on Concerta for at least 60 days and switch to authorized generic will be observed.
  Other Names: Methylphenidate
  Groups: Concerta to authorized generic (AG) formulation
Drug: Concerta EG formulation — This is an observational study. Participants who have been on Concerta for at least 60 days and switch to equivalent generic will be observed.
  Other Names: Methylphenidate
  Groups: Concerta to equivalent generic (EG) formulation

SUMMARY:
The primary purpose of this study is to identify whether, after adjustment for confounders via stratification on a propensity score and adjustment for calendar year, the combined endpoint consisting of #1 to #4 (1. switching back to Concerta, 2. changing the use of immediate release [IR] methylphenidate, 3. beginning a new attention deficit hyperactivity disorder [ADHD] medication, or 4. stopping both Concerta and the long acting [LA] methylphenidate {authorized generic [AG] methylphenidate or equivalent generic [EG] methylphenidate} that was begun on the index date), differs between participants who switch from branded Concerta to the EG formulations versus participants who switch from branded Concerta to the AG formulation.

DETAILED DESCRIPTION:
This is a retrospective cohort study based on a health claims database, the Truven Commercial Claims and Encounters (CCAE) database. Participants will enter the cohort when, after using Concerta continuously for at least 60 days after October 3, 2012, they receive a dispensing of the AG or EG formulation within 15 days of the end of the days of Concerta supplied. The date of that dispensing of the AG or EG formulation is the participants index date. This study will track various events, example, back-switches, and methylphenidate dose changes over time (the 60 days before the switch from Concerta to an AG or EG generic compared to the 60 days after that switch).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 6 to 65 years of age
* Have been in the database continuously for at least 183 days after June 1, 2012
* Have a diagnosis of attention deficit hyperactivity disorder (ADHD)
* Use Concerta (a brand of methylphenidate) for at least 60 days and receive a dispensing of the authorized generic (AG) or equivalent generic (EG) formulation within 15 days of the end of the days of Concerta supplied. The date of that dispensing of the EG or AG formulation is the participants index date
* Have an index date greater than or equal to (>=) Dec 1, 2012 and less than or equal to (<=) Dec 3, 2014, the former to reflect the fact that the EG preparation became available in December, 2012, and the latter to allow 60 days follow up <= Jan 31, 2015, which is the end date for the available data

Exclusion Criteria:

* Their age or sex is not specified in the database
* At any time after June 1, 2012 and before their index date they receive a diagnosis of Renal insufficiency or Hepatic insufficiency or Schizophrenia or Bipolar disorder or mania or Anxiety or Glaucoma or Tourettes's syndrome or Nervous tension or Narrowing of esophagus, stomach or intestine
* At any time from 183 days before they join the cohort to 60 days after their index date, they a) are diagnosed as pregnant; b) are dispensed any prescription medication commonly used to treat seizures or migraines c) are dispensed any antidepressant or antipsychotic medication
* At any time from 60 days before their index date to 60 days after their index date they a) Receive a dispensing of methylphenidate in any form other than a non-chewable tablet, example, if they receive methylphenidate as a patch, suspension, syrup, or chewable tablet b) Receive a dispensing of long acting (LA) methylphenidate other than Concerta, the AG formulation or an EG formulation
* Concerta is dispensed to the participant <= 3 days after the index date

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the Truven Commercial Claims and Encounters (CCAE) database who enroll in the study will have a confirmed diagnosis of ADHD and continuously used Concerta brand of methylphenidate for at least 60 days and receive a dispensing of the AG or EG formulation within 15 days of the end of the days of Concerta supplied.
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants Switching Back to Concerta | 60 Days after index date (the date when participant switches from Concerta to an AG or EG)
Number of Participants Changing the use of Immediate Release (IR) Methylphenidate | 60 Days after index date (the date when participant switches from Concerta to an AG or EG)
Number of Participants Starting a new Different Attention Deficit Hyperactivity Disorder (ADHD) Medication | 60 Days before index date (the date when participant switches from Concerta to an AG or EG)
Number of Participants Discontinuing the use of Both Concerta and the Study Drug to Which the Participant is Switched | 60 Days after index date (the date when participant switches from Concerta to an AG or EG)

SECONDARY OUTCOMES:
Number of Participants Changing the use of Immediate Release (IR) Methylphenidate | 60 Days before and after index (the date when participant switches from Concerta to an AG or EG)
Number of Participants Starting a new Different Attention Deficit Hyperactivity Disorder (ADHD) Medication | 60 Days after index date (the date when participant switches from Concerta to an AG or EG)
Number of Participants Changing an Established Methylphenidate | 60 Days after index date (the date when participant switches from Concerta to an AG or EG)
Number of Participants Having Outpatient Visits for ADHD | 60 days after the index date (the date when participant switches from Concerta to an AG or EG)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

REFERENCES:
- [Derived] Fife D, Cepeda MS, Baseman A, Richards H, Hu P, Starr HL, Sena AG. Medication changes after switching from CONCERTA(R) brand methylphenidate HCl to a generic long-acting formulation: A retrospective database study. PLoS One. 2018 Feb 28;13(2):e0193453. doi: 10.1371/journal.pone.0193453. eCollection 2018. PMID 29489906